CLINICAL TRIAL: NCT03142698
Title: Evaluation of 4 MRI Methods (PDFF 3, 6 and 11 Gradient Echoes and Spectroscopy) Compared to the Reference Method (Liver Biopsy) in Quantification of Hepatic Steatosis
Acronym: STEA-MRI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-317; 2016-A02065-46 (Other: 2016-A02065-46)
Record Dates: First submitted 2017-04-13; First posted 2017-05-05 (Actual); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Hepatic Steatosis; MRI; Liver Biopsy; Quantification
Keywords: hepatic steatosis; MRImaging
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hepatic steatosis (Experimental): Evaluation of different techniques in quantification of hepatic steatosis by MRImaging (PDFF 3, 6 and 11 gradient echoes and Spectroscopy) compared to the histological method (reference)
  Interventions: Procedure: Quantification of hepatic steatosis

INTERVENTIONS:
Procedure: Quantification of hepatic steatosis — Quantification of hepatic steatosis (histology, and in MRI)

SUMMARY:
Evaluation of 4 MRI methods (PDFF 3, 6 and 11 gradient echoes and Spectroscopy) compared to the reference method (liver biopsy) in quantification of hepatic steatosis

DETAILED DESCRIPTION:
Hepatic steatosis is an increasingly frequent pathology, which can lead to severe complications (Cirrhosis, Hepatocellular Carcinoma).

The poor quantification of steatosis by ultrasound or scanning and the invasiveness of the reference method (liver biopsy) make MRI a measurement tool of choice.

Recent techniques such as proton density measurement with several echoes or spectroscopy are increasingly used for the measurement of steatosis.

At the time of the development of therapeutics to reduce fatty liver disease, the use of MRI seems an interesting alternative for longitudinal follow-up in these patients.

Our study aims to ensure the reliability of these different MRI techniques for accurate quantification of liver steatosis and to compare them.

* Measurement and influence of hepatic fibrosis
* Measurement and influence of intrahepatic iron
* Influence of intercurrent liver disease
* Comparison of the fat measurement of the different hepatic segments
* Reproducibility by measurement of inter-observer concordance

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing hepatic biopsy (trans-parietal or trans-jugular) in the context of liver disease
* signature of written consent

Exclusion Criteria:

* Contra-indications to MRI
* Refusal of protocol
* underage patients and protected adults

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient - for each quantitative MRI variable studied - with the histological score of hepatic steatosis. | at day 1
  Correlation coefficient - for each quantitative MRI variable studied - with the histological score of hepatic steatosis.

SECONDARY OUTCOMES:
Measurement of intrahepatic iron | at day 1
Measurement of intrahepatic fibrosis | at day 1
Measurement of fat in different hepatic segments | at day 1
  (MRI )
Concordance between observers | at day 1
  (for MRI measurements)

CONTACTS AND LOCATIONS:
Overall Officials: Louis BOYER, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France